CLINICAL TRIAL: NCT06613763
Title: Pharmacokinetics of RAY1225 Following Administration to Subjects With Impaired Renal Function
Brief Title: A Study of RAY1225 in Participants With Impaired Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RAY1225-24-06
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-09

CONDITIONS: Kidney Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RAY1225 - Mild Renal Impairment (Experimental): RAY1225 3mg administered SC to participants with mild renal impairment.
  Interventions: Drug: RAY1225
- RAY1225 - Moderate Renal Impairment (Experimental): RAY1225 3mg administered SC to participants with moderate renal impairment.
  Interventions: Drug: RAY1225
- RAY1225 - Severe Renal Impairment (Experimental): RAY1225 3mg administered SC to participants with severe renal impairment.
  Interventions: Drug: RAY1225
- RAY1225 - Control (Experimental): RAY1225 3 milligrams (mg) administered subcutaneously (SC) to healthy participants with normal renal function.
  Interventions: Drug: RAY1225

INTERVENTIONS:
Drug: RAY1225 — Administered SC

SUMMARY:
The purpose of this study is to assess how fast RAY1225 gets into the blood stream and how long it takes the body to remove it in participants with impaired kidney function compared to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥18 to ≤28kg/m2 and total body weight >50 kg(male) or >40kg(female) at Screening (calculated as a function of measured height and weight according to the formula, BMI = kg / m2 where m2 is height in meters squared);
2. Ability to understand and willingness to sign a written informed consent form;

   Participants with normal renal function only:
3. Normal physical examination, vital signs, 12-lead ECG, Chest X-ray images (anteroposterior) and clinical laboratory values, or any abnormality that is non-clinically significant；
4. Glomerular filtration rate (GFR)≥ 90 mL/min and <130 mL/min ；
5. Age, BMI, and sex comparable to those of subjects of renal impairment；

   Participants with severe renal impairment only:
6. Diagnosis of CKD (any indicators of renal impairment or GFR < 60 mL/min/1.73 m2 for more than 3 months)；

Exclusion Criteria:

1. Participants with an allergic disposition (multiple drug and food allergies) or who, have known allergies to RAY1225 or related compounds;
2. Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2;
3. Participants who donated blood or bleeding profusely (> 400 mL) in the 3 months or donated blood or bleeding profusely (> 200 mL) in the 1 months;
4. Pregnant or lactating women, or women of childbearing age with a positive pregnancy test
5. Participants with serious infections, trauma, gastrointestinal surgery or other major surgical procedures within 4 weeks

   Participants with severe renal impairment only:
6. Participants with acute renal failure, or a kidney transplant history; or requiring renal dialysis during the study period;
7. Hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥ 160mm Hg or diastolic blood pressure ≥ 100mm Hg)
8. New York heart association (NYHA) class III or IV congestive heart failure
9. Alanine aminotransferase (ALT) ≥ 2×ULN, aspartate aminotransferase(AST) ≥ 2×ULN; Serum total bilirubin > 1.5×ULN;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of RAY1225 From Time Zero to T (AUC[0-t]) | Baseline through Day 43
PK: Maximum Concentration of RAY1225 | Baseline through Day 43

SECONDARY OUTCOMES:
Number and severity of participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events(SAE) | Baseline through Day 43

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China